CLINICAL TRIAL: NCT05178771
Title: The Efficacy of Application of Platelet-rich Fibrin on Periodontal Clinical Parameters and Gingival Crevicular Fluid Platelet-derived Growth Factor-BB and Periostin Levels
Brief Title: Efficacy of PRF Application on Clinical Parameters and GCF Platelet-derived Growth Factor-BB and Periostin Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Sarah Alrihaymee, Dentist, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRF effect on perio-parameters
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Periodontitis
Keywords: PRF; PDGF-BB; Periostin
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: A split-mouth procedure will be formed. Two quadrants in each participant will be selected; the sites will be divided into two groups: control site( will treat by ScRp only) and test sites( will treat by ScRp and PRF)
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed by coin toss method
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test site (Experimental): The test site will receive ScRp in addition to PRF
  Interventions: Other: Platelet rich fibrin
- control sites (No Intervention): The control site will be treated by ScRp only

INTERVENTIONS:
Other: Platelet rich fibrin — 1. Intravenous blood (obtained by venipuncture of the antecubital vein) will be collected in two 10-mL sterile tubes without any anticoagulants and will be immediately centrifuged at 3,000 revolutions (400 × g) per minute for 10 minutes.
  2. A structured fibrin clot in the middle of the tube, just between the red corpuscles (RBCs) at the bottom and the acellular plasma at the top, will be separated from the RBCs using sterile tweezers and scissors and transferred on a sterile PRF box.
  3. The PRF will be then brought to a thickness of 1 mm by gently compressing in PRF box. Standardized PRF pieces will be obtained by measuring by a periodontal probe and cutting into 3 × 5 mm dimensions.
  4. The PRF pieces will be inserted into the periodontal pockets by filling the pockets from the base up to the gingival margin. A modified gingivectomy knife, of which the tip is made blunt, will be used.
  The PRF volume will be calculated by recording how many pieces will be inserted.
  Arms: test site

SUMMARY:
Determine the efficacy of the non-invasive application of PRF on periodontal clinical parameters(pocket reduction) and the levels of PDGF-BB and Periostin in the gingival crevicular fluid.

DETAILED DESCRIPTION:
The adjunctive use of PRF with conventional ScRp may improve clinical healing, decrease tissue morbidities such as pain and discomfort, increase patient acceptance, reduce treatment time. Since PRF can be utilized as a safe, natural method to repair tissues at a low cost. Our aim is to evaluate the effectiveness of the non-invasive application of PRF as an adjunct to ScRp in patients with stage III grade B periodontitis through measurements of gingival crevicular fluid levels of PDGF-BB and Periostin before and after treatment and compare it with ScRp alone. A split-mouth procedure will be performed to reduce confounders as possible.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients.
* Patients with periodontitis.

Exclusion Criteria:

1. Medical history of systemic disease: diabetes, pregnancy, or lactation.
2. Previous periodontal treatment for the last 6 months
3. Grade II mobility
4. Smoker or alcoholic patient.
5. Teeth with untreated caries, endodontic lesions
6. Symptoms of recent acute illness e.g., COVID-19 will be excluded as well

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
clinical parameters | 4 weeks and 3 months
  measurements of pocket depth in millimeter at baseline and at the end of study

SECONDARY OUTCOMES:
PDGF-BB and periostin level in GCF | 4 weeks and 3 months
  Measurement of PDGF-BB and periostin level in GCF in baseline data and at the end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Babylon University, Hillah, Babel, Iraq

IPD SHARING:
Plan to Share IPD: No